CLINICAL TRIAL: NCT00963612
Title: Non-Invasive Prediction of Microvascular Invasion (MVI) in Hepatocellular Carcinoma (HCC) by Assessment of Tumor Oxygenation by Blood Oxygen Level-Dependent Magnetic Resonance Imaging (BOLD MRI)
Brief Title: Non-invasive Prediction of Microvascular Invasion in Hepatocellular Carcinoma by Blood-Oxygen-Level Dependent Magnetic Resonance Imaging (BOLD MRI)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: UHN09-0426-CE
Record Dates: First submitted 2009-08-07; First posted 2009-08-21 (Estimated); Last update posted 2017-10-02 (Actual); Status verified 2017-09

CONDITIONS: Hepatocellular Carcinoma
Keywords: Microvascular Invasion; Blood-Oxygen-Level Dependent Magnetic Resonance Imaging (BOLD MRI)
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single Arm (Other): In this project, there is only one study group which comprises of patients with Hepatocellular Carcinoma (HCC) who will undergo "Liver BOLD-MRI" before hepatic resection.
  Interventions: Procedure: BOLD MRI test

INTERVENTIONS:
Procedure: BOLD MRI test — Additional MR pulse sequence performed on BOLD MRI is expected to increase the regular scan time by an additional 5-10 minutes. No intravenous contrast is required for BOLD acquisition.

SUMMARY:
Liver resection and liver transplantation are the acceptable treatment of Hepatocellular Carcinoma (HCC). But the long-term survival is unsatisfactory as a result of high rate of intra and extra hepatic recurrences. Microvascular invasion (MVI) is the most significant risk factor affecting recurrence-free survival in patients following liver resection and liver transplantation. Tumor hypoxia (lack of adequate blood supply) is the single most important factor that predict MVI and post surgical prognosis.

Blood Oxygen Level Dependent (BOLD) MRI is a non-invasive diagnostic method of assessing tumor hypoxia by detecting signal changes secondary to changes in blood flow and oxygenation. BOLD MRI assessment of tumor hypoxia in HCC has never been correlated with pathological confirmation of MVI, the gold standard to assess MVI in HCC. In this study, the investigators propose to assess the ability of BOLD MRI to provide a discriminating quantitative threshold of intratumoral oxygenation predictive of MVI.

ELIGIBILITY:
Inclusion Criteria:

* Patients with known Hepatocellular Carcinoma;
* Scheduled to undergo liver resection or liver transplantation.

Exclusion Criteria:

* Estimated GFR (eGFR < 30 mL/min;
* MRI contrast allergy;
* General contraindications to MRI such as pacemaker, etc.;
* Prior tumor treatment such as transarterial chemoembolization or the tumor or radiofrequency ablation or chemoradiation;
* Pregnancy;
* Age less than 18 years.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2009-09; Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
To assess the ability of BOLD MRI to predict microvascular invasion in hepatocellular carcinoma via assessment of intratumoral oxygenation. | 18 months

SECONDARY OUTCOMES:
To identify a quantitative threshold tumor R2* value using BOLD MRI technique reasonably sensitive of predicting microvascular invasion in HCC pre-operatively. | 18 months

CONTACTS AND LOCATIONS:
Overall Officials: Kartik Jhaveri, MD, Principal Investigator — University Health Network, Toronto
Locations (1):
- University Health Network, Toronto, Ontario, Canada